CLINICAL TRIAL: NCT06279598
Title: PT-STRESS Study: A Two-phase RCT Aimed at Predicting Treatment Success and Dealing With Non-response in the Treatment of PTSD; by Alternating Between Two Trauma-focused Treatments (EMDR/PE) or by Switching to Interpersonal Therapy (IPT)
Brief Title: PT-STRESS Study: Predicting Treatment Success and Dealing With Non-response in the Treatment of PTSD
Acronym: PT-STRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Groningen (Other)
Collaborators: Dimence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversityGroningen
Record Dates: First submitted 2023-12-13; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Psychotherapy; Trauma; Prolonged Exposure; Eye Movement Desensitization Reprocessing; Interpersonal Psychotherapy; Trauma-focused Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing; Interpersonal Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial (RCT) conducted in two phases. Patients with PTSD will first be randomized to PE or EMDR in the first treatment phase. After this first phase of treatment, non-responders are re-randomized for a second phase of treatment. They receive either the alternative phase 1 trauma-focused psychotherapy or IPT as non-trauma-focused therapy for PTSD. In both phases (phase 1 and 2) the treatment lasts 8 weeks. Patients receive 14 sessions of 1 hour in 8 weeks.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolonged Exposure (Active Comparator): Intervention: Prolonged Exposure therapy, 14 sessions of 60 minutes in 8 weeks.
  Interventions: Behavioral: Prolonged Exposure therapy
- Eye Movement Desensitization Reprocessing (Active Comparator): Intervention: Eye Movement Desensitization Reprocessing (EMDR), 14 sessions of 60 minutes in 8 weeks.
  Interventions: Behavioral: Eye Movement Desensitization Reprocessing (EMDR)
- Interpersonal Psychotherapy (Experimental): Intervention: Interpersonal Psychotherapy (IPT), 14 sessions of 60 minutes in 8 weeks. In phase 2 of the study for treatment non-responders, IPT is studied as an alternative switching option compared to the switch of the aforementioned trauma-focused forms of psychotherapy.
  Interventions: Behavioral: Interpersonal Psychotherapy (IPT)

INTERVENTIONS:
Behavioral: Prolonged Exposure therapy — This concerns a form of psychotherapy for PTSD.
  Other Names: Trauma-focused CBT
  Arms: Prolonged Exposure
Behavioral: Eye Movement Desensitization Reprocessing (EMDR) — This concerns a form of psychotherapy for PTSD.
  Arms: Eye Movement Desensitization Reprocessing
Behavioral: Interpersonal Psychotherapy (IPT) — This concerns a form of psychotherapy for PTSD.
  Arms: Interpersonal Psychotherapy

SUMMARY:
The aim of this study is to increase understanding of the effectiveness and efficiency of psychological treatment for adult patients with posttraumatic stress disorder -PTSD- and to make it more personalized.

Key questions:

1. Which predictors of treatment success influence treatment outcome of patients with PTSD who receive the three psychotherapeutic treatments investigated in this study?
2. Which specific moderators can be identified with regard to the different psychotherapies (Eye Movement Desensitization and Reprocessing -EMDR-; Prolonged Exposure -PE-; and Interpersonal Psychotherapy -IPT- in the second phase)?
3. In patients with PTSD, does offering another proven effective form of trauma-focused psychotherapy (PE after EMDR, or EMDR after PE) improve symptoms following insufficient response to a first trauma-focused treatment?
4. Is switching from a trauma-focused therapy to a non-trauma-focused treatment (IPT) a more effective strategy for dealing with non-response to a first proven effective psychotherapeutic treatment compared to switching to another trauma-focused therapy?
5. Are there differences in treatment tolerance and differences in dropout rates between PE, EMDR and IPT?

Secondary goals:

* Investigating the extent to which therapist allegiance to a specific therapy method affects outcomes;
* Investigating whether the quality of therapy implementation or the treatment integrity ('adherence/ competence') affects treatment outcomes;
* Investigating how much the quality of the therapeutic alliance influences outcomes.

Participants receive treatment and will complete questionnaires. The study is conducted in two phases. Its aim is to compare two different trauma-focused treatments (EMDR and PE) for patients with PTSD to one another and with a nontrauma-focused psychotherapy (IPT) and to investigate possible predictors and moderators for treatment success. Patients will first be randomized to PE or EMDR in the first treatment phase. After this first phase, non-responders are re-randomized for a second phase of treatment. They receive either the alternative phase 1 trauma-focused psychotherapy or IPT as non-trauma-focused therapy. In phase 1 researchers will compare the PE and EMDR group to see which treatment is most effective for whom. In phase 2 researchers will compare the trauma-focused treatments (PE and EMDR group) with the nontrauma-focused treatment (IPT group) to see which treatment is most effective for whom.

DETAILED DESCRIPTION:
Background of the study:

The symptoms of posttraumatic stress disorder (PTSD) follow exposure to a traumatic event and are accompanied by significant functional limitations. PTSD is very common: a multinational study shows a lifetime prevalence of 3.9%. Effective treatment options exist for people with PTSD, with Eye Movement Desensitization and Reprocessing (EMDR) and Prolonged Exposure (PE; a specific form of trauma-focused Cognitive Behavioral Therapy, T-CBT) both listed as first-choice interventions in the Dutch standard of care for psychotrauma and stressor related disorders. About 40% of patients with PTSD do not benefit sufficiently from either of the aforementioned guideline treatments and about 18% of patients do not complete a trauma-focused treatment (treatment dropout). Knowledge about general predictors of treatment success in psychotherapy is limited, making it currently impossible to predict which patient will or will not benefit from which specific psychotherapeutic treatment (i.e., EMDR vs. PE). Little scientific knowledge exists about optimal follow-up treatment when patients insufficiently benefit from their initial treatment. For patients who drop out (e.g. from inability to tolerate exposure to traumatic memories) or do not benefit from exposure therapies, an alternative is to switch not to another proven effective trauma-focused intervention, but to a non-trauma-focused intervention. A suitable non-traumafocused treatment is Interpersonal Psychotherapy. Previous research suggests that IPT can be an effective first-line treatment option, but the effectiveness of IPT as a second treatment step for people with PTSD who have not responded to a trauma-focused psychotherapy has never been investigated. We hypothesize that IPT will yield greater symptom reduction and less dropout for patients with PTSD who do not respond to a course of trauma-focused psychotherapy compared to switching to another trauma-focused therapy.

Study population:

Subjects are recruited from Dimence, a mental health institution in the Netherlands. Subjects are recruited from patients who register for outpatient treatment within the Dimence division "Specialistic Diagnostics and Treatment" with a primary diagnosis of PTSD. It concerns adults between 18 and 65 years old, both men and women.

Intervention:

Half of initially non-responsive patients will be treated with the non-trauma-focused intervention interpersonal therapy (IPT) in phase 2 of the study. The first and second phases will offer the trauma-focused treatments Prolonged Exposure and EMDR.

* Interpersonal Psychotherapy (IPT) does not target the memories of a traumatic event but the interpersonal consequences of trauma, seeking to improve affective and interpersonal functioning that PTSD symptoms have disrupted. PTSD following a traumatic life event produces social withdrawal and a blunted, inhibited emotional life, disrupting interpersonal functioning. IPT helps benumbed patients recognize and tolerate their feelings so they can use them to handle their social environment, determine who is trustworthy, and mobilize protective social supports. IPT addresses patient emotions and their relationship to interpersonal interactions. As patients recognize their feelings, the therapist helps patients to name, normalize, and use their feelings rather than seeing them as an additional threat.
* In Prolonged Exposure, patients directly confront traumatic memories and cues and learn to expose themselves to terrifying but not dangerous stimuli to achieve habituation or extinction. The current study will use a protocol-based treatment of Cognitive Behavioral Therapy for PTSD that includes imaginal and in vivo exposure.
* In EMDR, patients are distracted from the traumatic memories by a dual attention task, usually using eye movements. This study will use a protocolled EMDR treatment for PTSD.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

Major adverse events are not expected as these have not been documented in previous studies. The greatest burden on subjects is completing the questionnaires necessary to answer the primary research questions. In phase 1, this totals approximately 10.5 hours (with baseline measurement the most extensive and subsequent weekly measurements); for patients treated for an additional 8 weeks in phase 2, completing the questionnaires takes approximately another 6 hours. A patient participating in both treatment phases therefore spends a total of approximately 16.5 hours completing assessments. The prescription of patients taking medication must be stable prior to the study, and then not changed during the study, unless necessary due to a crisis or serious side effects. Patients receive treatment sessions twice a week, which is relatively frequent compared to usual treatment, but research shows that dropout is lower with two weekly sessions. Study participation further assures patients that the treatments they receive are performed as intended by the therapy-developer because therapists receive supervision and checks are made to ensure treatment integrity.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 18 and 65 who were classified with a primary diagnosis of PTSD (based on the DSM-5 criteria).
* Adults who are willing to participate in the study (informed consent)

Exclusion Criteria:

* Insufficient proficiency in the Dutch language.
* Patients who cannot follow the treatment protocol (for example due to prolonged absence) are excluded from the study.
* Patients who use medication that is not stable. If properly set to the last prescribed medication by the doctor there will be advised to continue and referably not change the medication and its dose during treatment, unless necessary in connection with side effects, crisis, etc.
* Patients that already received an evidence-based form of trauma-oriented treatment for PTSD in the past year and for sufficient treatment duration, in accordance to the Dutch professional practice guidelines (reference: Akwa GGZ (2020, December 1). GGZ Standaarden. Psychotrauma- en stressorgerelateerde stoornissen. Retrieved September 29, 2022, from https://www.ggzstandaarden.nl/zorgstandaarden/psychotrauma-en-stressorgerelateerde-stoornissen/introductie).
* Patients with serious suicidality that requires acute intervention and structural addition of additional treatment interventions.
* Patients with an intellectual disability.
* Patients with a serious addiction as a comorbid problem.
* Patients with an acute mania or a psychotic state.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2031-05-20 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Measured every week for 8 weeks in phase 1 and measured every week of 8 weeks in phase 2 of the study.
  The primary outcome measure for the effectiveness of the treatment in both phases is symptom reduction (less burden of PTSD symptoms) measured with the PTSD checklist for the DSM-5 (PCL-5). The Dutch version of the PCL-5 will be used, the PCL-5 is administered at baseline and repeated weekly. The PCL-5 is a self-report questionnaire of 20 items about the DSM-5 symptoms of PTSD. This measure will be used to monitor symptom change during and after treatment in both phases of the study.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Measured at baseline, at the end of treatment in phase 1 (= after 8 weeks) and at the end of the treatment in phase 2 (= after 16 weeks = end of the study).
  The Dutch version of the CAPS-5 will be used as it is "the gold standard" in PTSD assessment. The CAPS-5 is a 30-item structured clinical interview that we will use, among other things, to determine the current (past month) diagnosis of PTSD and to assess improvement in symptoms since a previous CAPS administration.
International Trauma Questionnaire (ITQ) | Measured at baseline, at the end of treatment in phase 1 (= after 8 weeks) and at the end of the treatment in phase 2 (= after 16 weeks = end of the study).
  The Dutch version of the ITQ will be used: "Internationale Trauma Vragenlijst" (ITV). The International Trauma Questionnaire (ITQ) is a self-report questionnaire consisting of 18 items that measures complex PTSD (C-PTSD) symptoms according to the diagnostic criteria of the 11th revision of the International Classification of Diseases (ICD-11; World Health Organization).
Hospital Anxiety and Depression Scale (HADS) | Measured every week for 8 weeks in phase 1 and measured every week of 8 weeks in phase 2 of the study.
  The Dutch version of the HADS will be used. The Hospital Anxiety and Depression Scale is a 14-item self-report questionnaire and can be used to measure levels of anxiety and depression.
Mental Health Continuum Short Form (MHC-SF) | Measured at baseline, at the end of treatment in phase 1 (= after 8 weeks) and at the end of the treatment in phase 2 (= after 16 weeks = end of the study).
  The Dutch version of the MHC-SF will be used: the Dutch short-form Mental Health Continuum. The MHC-SF comprises 40 items that measure emotional well-being, psychological well-being and social well-being.
Positive and Negative Experiences of Psychotherapy questionnaire (PNEP) | Measured at baseline, at the end of treatment in phase 1 (= after 8 weeks) and at the end of the treatment in phase 2 (= after 16 weeks = end of the study).
  The Dutch version of the self-report questionnaire Positive and Negative Effects of Psychological Treatment (PNEP) will be used to assess both positive and possibly unfavorable and adverse events in psychological treatments. The Dutch questionnaire consists of 3 questions and 71 items.

OTHER OUTCOMES:
Age | Measured at baseline.
  We are investigating generic predictors of treatment success and specific moderators based on the scientific literature. Further, we have added several instruments to match those that Wibbelink et al. (2021) use in their research in order to be able to collaborate in future data analyses (PAI analysis).
  The first demographic variable is age.
Gender | Measured at baseline.
  We ask about gender.
Education | Measured at baseline.
  We ask about the level of education.
Employment | Measured at baseline.
  We ask about employment status.
Marital status | Measured at baseline.
  We ask about marital status.
Ethnicity/race | Measured at baseline.
  We ask about ethnicity/race.
Medication use | Measured at baseline.
  We ask about medication use.
Treatment history | Measured at baseline.
  We ask about treatment history.
Mini-Schedules for Clinical Assessment in Neuropsychiatry (mini-SCAN) | Measured at baseline.
  The Mini-Schedules for Clinical Assessment in Neuropsychiatry is a shortened version of the SCAN 2.1 developed by the World Health Organization (WHO). The Mini-SCAN is a semi-structured diagnostic interview that determines the most common DSM-5 (formerly DSM-IV Axis I) diagnoses using a diagnostic algorithm. The instrument is administered at baseline in the study to determine comorbidity of other disorders with PTSD, including depression, anxiety, and substance use disorders.
Life Events Checklist for DSM-5 (LEC-5) | Measured at baseline.
  The Life Events Checklist for DSM-5 (LEC-5) is often used as a standard lead-in to the CAPS-5 to determine Criterion A validity. The LEC-5 comprises 17 items.
The Childhood Trauma Questionnaire-Short Form (CTQ-SF) | Measured at baseline.
  The Childhood Trauma Questionnaire-Short Form (CTQ-SF) will be administered at baseline to assess the severity of five types of child abuse: emotional abuse, physical abuse, sexual abuse, emotional neglect and physical neglect. The CTQ-SF consists of 28 items.
Symptom Checklist-90 (SCL-90), Hostility subscale | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  The "Hostility" subscale of the Symptom Checklist-90-Revised (SCL-90-R) will be used to measure anger. This subscale of the SCL-90-R consists of 6 items rated on a 5-point Likert scale ranging from 0 ('not at all') to 4 ('extremely') and assesses anger-related thoughts, feelings, and actions.
Experiences in Close Relationships-Relationship Structures (ECR-RS) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  General attachment style will be measured using the Experiences in Close Relationships-Relationship Structures questionnaire (ECR-RS). The ECR-RS comprises 9 items rated on a 7-point Likert scale ranging from 1 ('completely disagree') to 7 ('completely agree). The ECR-RS measures attachment-related avoidance and attachment-related anxiety.
The Brief Experiental Avoidance Questionnaire (BEAQ) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  The Brief Experiential Avoidance Questionnaire (BEAQ) will be used to measure experiential avoidance. The BEAQ measures six different domains: behavioral avoidance, fear aversion, suppression, procrastination, repression/denial and distress endurance. The BEAQ comprises 15 items rated on a 6-point Likert scale from 1 ('strongly disagree') to 6 ('totally agree').
Improving Access to Psychological Therapies (IAPT) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  Social problems (including housing problems, unemployment, social isolation) will be assessed with a list of social problems derived from the Improving Access to Psychological Therapies (IAPT) program.
Posttraumatic Cognitions Inventory (PTCI) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  The Posttraumatic Cognitions Inventory (PTCI) is a questionnaire consisting of 33 items that assess trauma-related cognitions measured in three domains: negative cognitions about oneself, negative cognitions about the world, and self-blame.
Trauma Related Guilt Inventory (TRGI) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  The Trauma Related Guilt Inventory (TRGI) will be administered to measure feelings of guilt related to the trauma. The questionnaire consists of 32 items rated on a 5-point Likert scale.
Trauma Related Shame Iventory (TRSI) | Measured at baseline and at the end of treatment in phase 1 (= after 8 weeks).
  A Dutch translation of the Trauma Related Shame Inventory (TRSI) will be administered to measure shame. Shame is defined in the TRSI as a negative and painful self-evaluation in the traumatic context and a tendency to withdraw and hide from others. The questionnaire comprises 24 items rated on a 4-point Likert scale from 1 ('not true for me') to 4 ('completely true for me').
Working Alliance Questionnaire shortened version (WAV-12) | Measured every week for 8 weeks in phase 1 and measured every week of 8 weeks in phase 2 of the study.
  The therapeutic relationship will be measured with the Working Alliance Questionnaire - shortened version (WAV-12). The WAV-12 is derived from the WAV-36, the Dutch translation from the Working Alliance Inventory (WAI). The questionnaire measures the bond between patient and therapist, agreement on the goals of treatment and agreement on the tasks in therapy. The WAV-12 consists of 12 items rated on a 5-point Likert scale from 1 ('rarely or never') to 5 ('always').
Expectancy rating (patients and therapists) | Measured at baseline.
  An 'expectancy rating' will be used to assess the expectations of patiens and practitioners of the treatment methods offered in the study (Prolonged Exposure, EMDR and IPT).This expectancy rating is administered at baseline and comprises 3 items (one about Prolonged Exposure, one about EMDR and one about IPT) in which patients and practitioners assess the expectation that the therapy will help the patient on scale from 0 ('not at all') to 100 ('maximum').

CONTACTS AND LOCATIONS:
Overall Officials: Maarten K van Dijk, PhD, Principal Investigator — Dimence
Locations (1):
- Dimence, Deventer, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boeschoten MA, Van der Aa N, Bakker A, Ter Heide FJJ, Hoofwijk MC, Jongedijk RA, Van Minnen A, Elzinga BM, Olff M. Development and Evaluation of the Dutch Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Eur J Psychotraumatol. 2018 Nov 22;9(1):1546085. doi: 10.1080/20008198.2018.1546085. eCollection 2018. PMID 30510643
- [Background] Loerinc AG, Meuret AE, Twohig MP, Rosenfield D, Bluett EJ, Craske MG. Response rates for CBT for anxiety disorders: Need for standardized criteria. Clin Psychol Rev. 2015 Dec;42:72-82. doi: 10.1016/j.cpr.2015.08.004. Epub 2015 Aug 14. PMID 26319194
- [Background] Mavranezouli I, Megnin-Viggars O, Daly C, Dias S, Welton NJ, Stockton S, Bhutani G, Grey N, Leach J, Greenberg N, Katona C, El-Leithy S, Pilling S. Psychological treatments for post-traumatic stress disorder in adults: a network meta-analysis. Psychol Med. 2020 Mar;50(4):542-555. doi: 10.1017/S0033291720000070. Epub 2020 Feb 17. PMID 32063234
- [Background] Coventry PA, Meader N, Melton H, Temple M, Dale H, Wright K, Cloitre M, Karatzias T, Bisson J, Roberts NP, Brown JVE, Barbui C, Churchill R, Lovell K, McMillan D, Gilbody S. Psychological and pharmacological interventions for posttraumatic stress disorder and comorbid mental health problems following complex traumatic events: Systematic review and component network meta-analysis. PLoS Med. 2020 Aug 19;17(8):e1003262. doi: 10.1371/journal.pmed.1003262. eCollection 2020 Aug. PMID 32813696
- [Background] Markowitz, J. C. (2021). Interpersoonlijke psychotherapie bij posttraumatische stressstoornis: Een nieuwe vorm van traumabehandeling (1e druk). Bohn Stafleu van Loghum.
- [Background] Bleiberg KL, Markowitz JC. Interpersonal Psychotherapy for PTSD: Treating Trauma without Exposure. J Psychother Integr. 2019 Mar;29(1):15-22. doi: 10.1037/int0000113. PMID 31534308
- [Background] Levinson DB, Halverson TF, Wilson SM, Fu R. Less dropout from prolonged exposure sessions prescribed at least twice weekly: A meta-analysis and systematic review of randomized controlled trials. J Trauma Stress. 2022 Aug;35(4):1047-1059. doi: 10.1002/jts.22822. Epub 2022 Mar 12. PMID 35278229
- [Background] Hoppen TH, Lindemann AS, Morina N. Safety of psychological interventions for adult post-traumatic stress disorder: meta-analysis on the incidence and relative risk of deterioration, adverse events and serious adverse events. Br J Psychiatry. 2022 Aug 12:1-10. doi: 10.1192/bjp.2022.111. Online ahead of print. PMID 35959698
- [Background] De Jongh, A., & Ten Broeke, E. (2019). Handboek EMDR. Een geprotocolleerde behandelmethode voor de gevolgen van psychotrauma (7e editie). Pearson.
- [Background] Van Minnen, A., & Arntz, A. (2017). Protocollaire behandeling van patiënten met posttraumatische-stressstoornis (PTSS). Imaginaire exposure en exposure in vivo. In G. Keijsers, A. Van Minnen, M. Verbraak, K. Hoogduin, P. Emmelkamp (Reds), Protocollaire behandelingen voor volwassenen met psychische klachten deel 1 (pp. 311-352). Boom.
- [Background] Koenen KC, Ratanatharathorn A, Ng L, McLaughlin KA, Bromet EJ, Stein DJ, Karam EG, Meron Ruscio A, Benjet C, Scott K, Atwoli L, Petukhova M, Lim CCW, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Bunting B, Ciutan M, de Girolamo G, Degenhardt L, Gureje O, Haro JM, Huang Y, Kawakami N, Lee S, Navarro-Mateu F, Pennell BE, Piazza M, Sampson N, Ten Have M, Torres Y, Viana MC, Williams D, Xavier M, Kessler RC. Posttraumatic stress disorder in the World Mental Health Surveys. Psychol Med. 2017 Oct;47(13):2260-2274. doi: 10.1017/S0033291717000708. Epub 2017 Apr 7. PMID 28385165
- [Background] Boeschoten, M. A., Bakker, A., Jongedijk, R. A., & Olff, M. (2014). PTSD Checklist for DSM-5 (PCL-5). Scale available from Stichting Centrum '45, Arq Psychotrauma Expert Groep. https://www.psychotraumadiagnostics.centrum45.nl/nl/ptss.nl
- [Background] Weathers, F. W., Blake, D. D., Schnurr, P. P., Kaloupek, D. G., Marx, B. P., & Keane, T. M. (2013). The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD. https://www.ptsd.va.gov
- [Background] Nienhuis, F. J., & Giel, R. (2000). Mini-SCAN voor klinisch gebruik. Swets & Zeitlinger.
- [Background] Eidhof, M., Ter Heide, F.J.J., Boeschoten, M.A., Olff, M. (2018). Internationale Trauma Vragenlijst: zelfrapportage vragenlijst voor ICD-11 PTSS en CPTSS. Nederlandstalige versie. Arq Psychotrauma Expert Groep. Scale available from http://www.psychotraumadiagnostics.centrum45.nl
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Lamers SM, Westerhof GJ, Bohlmeijer ET, ten Klooster PM, Keyes CL. Evaluating the psychometric properties of the Mental Health Continuum-Short Form (MHC-SF). J Clin Psychol. 2011 Jan;67(1):99-110. doi: 10.1002/jclp.20741. PMID 20973032
- [Background] Dandachi-FitzGerald, B., Houben, S. T. L., Broers, N. J., & Merckelbach, H. (2023). The Positive and Negative Experiences of Psychotherapy Questionnaire (PNEP): first psychometric findings of a new instrument for monitoring clients' experiences [Ongepubliceerd manuscript]. Afdeling Klinische Psychologie, Universiteit Maastricht; Faculteit Psychologie, Open Universiteit Heerlen.
- [Background] Weathers, F. W., Blake, D. D., Schnurr, P. P., Kaloupek, D. G., Marx, B. P., & Keane, T. M. (2013). The Life Events Checklist for DSM-5 (LEC-5). Instrument available from the National Center for PTSD. https://www.ptsd.va.gov
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Fraley RC, Heffernan ME, Vicary AM, Brumbaugh CC. The Experiences in Close Relationships-Relationship Structures questionnaire: a method for assessing attachment orientations across relationships. Psychol Assess. 2011 Sep;23(3):615-25. doi: 10.1037/a0022898. PMID 21443364
- [Background] Derogatis, L.R. (1977). SCL-90-R Symptom Checklist-90-R Administration, Scoring, and Procedures Manual. PsychCorp.
- [Background] Gamez W, Chmielewski M, Kotov R, Ruggero C, Suzuki N, Watson D. The brief experiential avoidance questionnaire: development and initial validation. Psychol Assess. 2014 Mar;26(1):35-45. doi: 10.1037/a0034473. Epub 2013 Sep 23. PMID 24059474
- [Background] Stinckens, N., Ulburghs, A., & Claes, L. (2009). De werkalliantie als sleutelelement in het therapiegebeuren: meting met behulp van de WAV-12, de Nederlandstalige verkorte versie van de Working Alliance Inventory. Tijdschrift Klinische Psychologie, 39(1), 44-60.
- [Background] Vervaecke, C.A.G., & Vertommen H. (1996). De Werk Alliantie Vragenlijst (wav). Gedragstherapie, 2, 139-144.
- [Background] Clark DM. Implementing NICE guidelines for the psychological treatment of depression and anxiety disorders: the IAPT experience. Int Rev Psychiatry. 2011 Aug;23(4):318-27. doi: 10.3109/09540261.2011.606803. PMID 22026487
- [Background] Foa, E. B., Ehlers, A., Clark, D. M., Tolin, D. F., & Orsillo, S. M. (1999). The Posttraumatic Cognitions Inventory (PTCI): development and validation. Psychological Assessment, 11(3), 303-314. https://doi-org.proxy-ub.rug.nl/10.1037/1040-3590.11.3.303
- [Background] Kubany, E. S., Haynes, S. N., Abueg, F. R., Manke, F. P., Brennan, J. M., & Stahura, C. (1996). Development and validation of the Trauma-Related Guilt Inventory (TRGI). Psychological Assessment, 8(4), 428-444. https://doi-org.proxy-ub.rug.nl/10.1037/1040-3590.8.4.428
- [Background] Øktedalen, T., Hagtvet, K. A., Hoffart, A., Langkaas, T. F., & Smucker, M. (2014). The Trauma Related Shame Inventory: Measuring trauma-related shame among patients with PTSD. Journal of Psychopathology and Behavioral Assessment, 36(4), 600-615. https://doi-org.proxy-ub.rug.nl/10.1007/s10862-014-9422-5
- [Background] Horvath, A. O., & Greenberg, L. S. (1989). Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology, 36(2), 223-233. https://doi.org/10.1037/0022-0167.36.2.223
- [Background] Wibbelink CJM, Lee CW, Bachrach N, Dominguez SK, Ehring T, van Es SM, Fassbinder E, Kohne S, Mascini M, Meewisse ML, Menninga S, Morina N, Rameckers SA, Thomaes K, Walton CJ, Wigard IG, Arntz A. The effect of twice-weekly versus once-weekly sessions of either imagery rescripting or eye movement desensitization and reprocessing for adults with PTSD from childhood trauma (IREM-Freq): a study protocol for an international randomized clinical trial. Trials. 2021 Nov 27;22(1):848. doi: 10.1186/s13063-021-05712-9. PMID 34838102